CLINICAL TRIAL: NCT01675310
Title: EFFECTIVITY OF MEDICAL NUTRITION THERAPY PLUS TRANSGESTATIONAL METFORMIN FOR PREVENTING THE INCIDENCE OF GESTATIONAL DIABETES MELLITUS IN HIGH RISK MEXICAN WOMEN.
Brief Title: Medical Nutrition Therapy Plus Transgestational Metformin For Preventing Gestational Diabetes In High Risk Mexican Women
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Instituto Nacional de Perinatologia Isidro Espinosa de los Reyes (Other Government)
Collaborators: National Council of Science and Technology, Mexico (Other)
Responsible Party: Principal Investigator, ENRIQUE REYES-Munoz MD, Clinical Reseach, Instituto Nacional de Perinatologia Isidro Espinosa de los Reyes
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Conacyt 151819; INPer (Mexico) (Registry Identifier: 21225042101)
Record Dates: First submitted 2012-08-27; First posted 2012-08-29 (Estimated); Last update posted 2015-03-25 (Estimated); Status verified 2015-03

CONDITIONS: Pregestational Obesity (BMI > 27kg/m2); History of Polycystic Ovary Syndrome
Keywords: obesity, polycystic ovary syndrome, gestational diabetes
MeSH Terms: conditions — Obesity; Polycystic Ovary Syndrome; Diabetes, Gestational | interventions — Nutrition Therapy; Metformin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- medical nutrition therapy + metformin (Experimental): medical nutrition therapy plus trans-gestational metformin (850mg 2 times day)
  Interventions: Drug: medical nutrition therapy + metformin
- medical nutrition therapy (Active Comparator): medical nutrition therapy without trans-gestational metformin
  Interventions: Behavioral: Medical nutrition therapy

INTERVENTIONS:
Drug: medical nutrition therapy + metformin
  Arms: medical nutrition therapy + metformin
Behavioral: Medical nutrition therapy — medical nutrition therapy
  Arms: medical nutrition therapy

SUMMARY:
Gestational diabetes mellitus is one of the most frequent complications of pregnancy, that affect between 1 to 14% of population around the world.

There is a few studies to prevent gestational diabetes mellitus in high risk women as Mexican population.

Metformin has been used during pregnancy in women with gestational diabetes and women with polycystic ovary syndrome, with acceptable security for mother and fetus.

Metformin decrease the insulin resistance and weight gain, we believe that metformin may be decrease the risk of gestational diabetes mellitus in high risk women.

ELIGIBILITY:
Inclusion Criteria:

* Mexican women with pregnancy < 16 weeks of gestation, normal oral glucose tolerance 75g-2h test and 3 or more criteria:

  1. Body mass index > 27 kg/m2
  2. Maternal age >25
  3. History of infertility with polycystic ovary syndrome
  4. History of macrosomic newborn (Weight >4000g)
  5. History of diabetes mellitus in first or second degree.
  6. History of gestational diabetes in previous pregnancy

Exclusion Criteria:

* Any form of pregestational diabetes
* Fasting glucose > 126 mg/dL at first prenatal visit.
* seric creatinine > 1.5 mg/dL
* Hyperthyroidism
* Heart disease
* Hepatic disease
* Renal diseases
* Epilepsy
* Lupus
* Chronic hypertension.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 90 (Actual)
Dates: Start 2012-01; Primary Completion 2014-12 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Gestational diabetes mellitus | 27-28 weeks of gestation
  oral glucose tolerance test

SECONDARY OUTCOMES:
insulin resistance | At birth
  measure of insulin resistance by HOMA-IR, sample of umbilical cord

CONTACTS AND LOCATIONS:
Overall Officials: Enrique Reyes-Muñoz, PhD, Principal Investigator — National Institute of Perinatology, Mexico City
Locations (1):
- National Institute of Perinatology, México, State of Mexico, Mexico

REFERENCES:
- [Derived] Perichart-Perera O, Mier-Cabrera J, Flores-Robles CM, Martinez-Cruz N, Arce-Sanchez L, Alvarado-Maldonado IN, Montoya-Estrada A, Romo-Yanez J, Rodriguez-Cano AM, Estrada-Gutierrez G, Espino Y Sosa S, Guzman-Huerta M, Ayala-Yanez R, Reyes-Munoz E. Intensive Medical Nutrition Therapy Alone or with Added Metformin to Prevent Gestational Diabetes Mellitus among High-Risk Mexican Women: A Randomized Clinical Trial. Nutrients. 2021 Dec 24;14(1):62. doi: 10.3390/nu14010062. PMID 35010938
- See also: Medical Nutrition Therapy Plus Metformin for Preventing Gestational Diabetes Among High-Risk Women. — http://journals.lww.com/greenjournal/Abstract/2014/05001/Medical_Nutrition_Therapy_Plus_Metformin_for.346.aspx